**Title of Research Study:** Reducing cervical cancer screening disparities through a primary care based HPV self-sampling intervention (Isbaar Project)

## **Investigator Team Contact Information:**

For questions about research appointments, the research study, research results, or other concerns, call the study team at:

Investigator Name: Rebekah Pratt, PhD Departmental Affiliation: Family Medicine

and Community Health

Phone Number: 612-625-1196 Email Address: rjpratt@umn.edu Study Staff: Christina Bliss Barsness Phone Number: 612-625-7179 Email Address: isbaar@umn.edu

If your doctor is also the person responsible for this research study, please note that s/he is interested in both your clinical care and the conduct of this research study. You have the right to discuss this study with another person who is not part of the research team before deciding whether to participate in the research.

**Supported By:** This research is supported by the National Cancer Institute.

# **Key Information About This Research Study**

The following is a short summary to help you decide whether or not to be a part of this research study. More detailed information is listed later on in this form.

#### What is research?

Doctors and investigators are committed to your care and safety. There are important differences between research and treatment plans:

- The goal of research is to learn new things in order to help groups of people in the future.
   Investigators learn things by following the same plan with a number of participants, so they do not usually make changes to the plan for individual research participants. You, as an individual, may or may not be helped by volunteering for a research study.
- The goal of clinical care is to help you get better or to improve your quality of life. Doctors can make changes to your clinical care plan as needed.

Research and clinical care are often combined. One purpose of this informed consent document is to provide you clear information about the specific research activities of this study.

#### Why am I being asked to take part in this research study?

We are asking you to take part in a follow-up interview for this research study because you previously had a self-sampled HPV test for an earlier phase of this study.

#### What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.


TEMPLATE LAST REVISED: 11/1/2021
Version Date: 7 January 2025

## Why is this research being done?

Our goal is to find out if offering HPV self-sampling tests will increase rates of cervical cancer screening for patients at primary care clinics. While this study has a primary focus on Somali patients who did the HPV self-sampling test, we will be conducting follow-up interviews with any patient who did the self-sample HPV test to learn more about their views and experiences with HPV self-sampling, getting a broad range of perspectives. We will use the information gathered from these interviews to identify strategies to better implement HPV self-sampling as a cervical cancer screening option in primary care clinics.

## How long will the research last?

We expect that you will be in this research study for one interview that will last approximately 30 minutes.

## What will I need to do to participate?

You will be asked to participate in an interview in an interview about your experience with HPV self-sampling.

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"

#### Is there any way that being in this study could be bad for me?

You may feel uncomfortable while talking about your experience with HPV self-sampling or other methods of cervical cancer screening. Research staff will be available to talk through any feelings of discomfort or concerns you may have.

A risk of participating in this study is that confidential information about you may be accidentally disclosed. However, this is an extremely unlikely event considering all the protective measures and precautions taken by the University and the research team.

### Will being in this study help me in any way?

There are no benefits to you from your taking part in this research. We cannot promise any benefits to others from your taking part in this research. However, possible benefits to others include improving and expanding access to cervical cancer screening options in the future.

#### What happens if I do not want to be in this research?

There are no known alternatives, other than deciding not to participate in this research study.

# **Detailed Information About This Research Study**

The following is more detailed information about this study in addition to the information listed above.

#### How many people will be studied?

We expect about 30 people will participate in the follow-up interviews for this research study.

## What happens if I say "Yes, I want to be in this research"?

You will be asked to review and sign this Consent Form and HIPAA Authorization either in-person or remotely via Zoom. Once you have signed this form and agreed to participate, research staff will review your medical record to verify that you are eligible to participate and confirm that you have completed any follow-up tests or treatment, depending on your results. You will receive multiple appointment reminders before your interview, based on your preferred method of contact.


TEMPLATE LAST REVISED: 11/1/2021
Version Date: 7 January 2025

The interview can take place in-person or remotely via Zoom or over the phone. You will be asked questions about your views on HPV self-sampling, your experience with HPV self-sampling, and the follow-up care you received if your test was positive. The interview will be audio recorded.

### What happens if I say "Yes", but I change my mind later?

If you take part in this research study, and want to leave, you should tell us. Your choice not to be in this study will not negatively affect your right to any present or future medical care, your academic standing as a student, or your present or future employment.

If you stop being in the research, information about you that has already been collected may not be removed from the study database.

### Will it cost me anything to participate in this research study?

Taking part in this research study will not lead to any costs to you.

# What happens to the information collected for the research, including my health information?

We try to limit the use and sharing of your information, including research study records, any medical records and any other information about you, to people who have a need for this information. But we cannot promise complete confidentiality.

#### **Overview**

If you participate in this study, your information, including your health information, will be used and shared for purposes of conducting this research. As described later in this Consent Form, your information may also be used and shared for publishing and presenting the research results, future research, and any optional elements of the research you agree to in this Consent Form, which may include creating audio and video recordings of you. If you sign this Consent Form, you are giving us permission to use and share your health information for these purposes, and if we are using your medical records, you are giving permission to any health care providers who are treating you to share your medical records with us.

#### What health information will be made available?

Health information about you to be used and shared for the research includes those items checked by the research team below:

☑ Your medical records, which may include records from hospital and clinic visits, emergency room visits, immunizations, medical history and physical exams, medications, images and imaging reports, progress notes, psychological tests, EEG/EKG/ECHO reports, lab and pathology reports, dental records and/or financial records. These records may be used and shared for as long as this research continues.

☑ Information collected as part of this research study, including research procedures, research visits, and any optional elements of the research you agree to, all as described in this Consent Form. This information might not be part of your medical record, and may include things like responses to surveys and questionnaires, and information collected during research visits described in this Consent Form.

What about more sensitive health information?

 TEMPLATE LAST REVISED: 11/1/2021 Version Date: 7 January 2025

Some health information is so sensitive that it requires your specific permission. If this research study requires any of this sensitive information, the boxes below will be marked and you will be asked to initial to permit this information to be made available to the research team to use and share as described in this Consent Form.

My drug & alcohol abuse, diagnosis & treatment records \_\_\_\_\_ (initial)

☐ My HIV/AIDS testing records \_\_\_\_\_\_ (initial)
 ☐ My genetic testing records \_\_\_\_\_\_ (initial)
 ☐ My mental health diagnosis/treatment records \_\_\_\_\_ (initial)
 ☐ My sickle cell anemia records \_\_\_\_\_ (initial)

Who will access and use my health information?

If you agree to participate in this study, your information will be shared with:

- The University of Minnesota research team and any institutions or individuals collaborating on the research with us;
  - Our collaborators at the University of Washington
  - Your medical service provider (Smiley's Family Medicine Clinic, People's Center Clinic, or the Community-University Health Care Center [CUHCC])
- Others at the University of Minnesota and M Health/Fairview who provide support for the
  research or who oversee research (such as the Institutional Review Board or IRB which is the
  committee that provides ethical and regulatory oversight of research at the University, systems
  administrators and other technical and/or administrative support personnel, compliance and
  audit professionals (Such as the Quality Assurance Program of the Human Research Protection
  Program (HRPP)), individuals involved in processing any compensation you may receive for your
  participation, and others);
- The research sponsor(s), any affiliates, partners or agents of the sponsor(s) involved in the research, organizations funding the research, and any affiliates, partners or agents of the funding organization(s) involved in the research;
- Organizations who provide accreditation and oversight for research and the research team, and others authorized by law to review the quality and safety of the research (such as U.S. government agencies like the Food and Drug Administration, the Office of Human Research Protections, the Office of Research Integrity, or government agencies in other countries); and
- Organizations that process any payments that may be made to you for participating in this study, and any other individuals or organizations specifically identified in this Consent Form.

#### Additional sharing of your information for mandatory reporting

If we learn about any of the following, we may be required or permitted by law or policy to report this information to authorities:

- Current or ongoing child or vulnerable adult abuse or neglect;
- Communicable, infectious or other diseases required to be reported under Minnesota's

 TEMPLATE LAST REVISED: 11/1/2021 Version Date: 7 January 2025

Reportable Disease Rule;

- Certain wounds or conditions required to be reported under other state or federal law; or
- Excessive use of alcohol or use of controlled substances for non-medical reasons during pregnancy.

#### How will my information be used in publications and presentations?

We may publish the results of this research in scientific, medical, academic or other journals or reports, or present the results at conferences. Information that makes it easy to identify you (such as your name and contact information, SSN and medical records number) will not be part of any publication or presentation. If you have an extremely unique or rare condition that is not shared by many others, it is possible that some people may be able to determine your identity even without these identifiers.

## What will be done with my data when this study is over?

Your data will not be used for any future research after this study is complete.

# Do I have to sign this Consent Form and give my permission to make my information, including my health information, available for use and sharing?

No, you do not have to sign this Consent Form. But if you do not sign, you will not be able to participate in this research study. Treatment available outside of the study, payment for such treatment, enrollment in health insurance plans and eligibility for benefits will not be impacted by your decision about signing this Consent Form.

#### Does my permission for making my health information available for use and sharing ever expire?

No, there is no expiration date.

#### May I cancel my permission for making my health information available for use and sharing?

Yes. You may cancel your permission at any time by writing to the researcher at the address on the first page of this Consent Form. If you cancel your permission, you will no longer be in the research study. You may also want to ask someone on the research team in canceling will affect any research related medical treatment. If you cancel your permission, any health information about you that was already used and shared may continue to be used and shared for the research study and any optional elements of the study to which you agree in this Consent Form.

#### What happens to my health information after it is shared with others?

When we share your information with others as described in this Consent Form, privacy laws may no longer protect your information and there may be further sharing of your information.

#### Will I be able to look at my records?

It is possible that the research team may not allow you to see the information collected for this study. However, you may access any information placed in your medical records after the study is complete.

#### **Certificate of Confidentiality**

To help protect your privacy, the National Institutes of Health has granted a Certificate of Confidentiality. The researchers can use this Certificate legally to refuse to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings,

 TEMPLATE LAST REVISED: 11/1/2021 Version Date: 7 January 2025

for example, if there is a court subpoena. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below.

The Certificate does not prevent a researcher from reporting information learned in research when required by other state or federal laws, such as mandatory reports to local health authorities for abuse or neglect of children/vulnerable adults, or information to the Food and Drug Administration (FDA) when required in an FDA audit. However, the Certificate limits the researcher from disclosing such information in follow up civil, criminal, legislative or administrative legal proceedings if the information was created or compiled for purposes of the research.

You also should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, medical care provider, or other person obtains your written consent to receive research information, then the researchers will not use the Certificate to withhold that information.

## Will anyone besides the study team be at my consent meeting?

You may be asked by the study team for your permission for an auditor to observe your consent meeting. Observing the consent meeting is one way that the University of Minnesota makes sure that your rights as a research participant are protected. The auditor is there to observe the consent meeting, which will be carried out by the people on the study team. The auditor will not document any personal (e.g. name, date of birth) or confidential information about you. The auditor will not observe your consent meeting without your permission ahead of time.

#### Whom do I contact if I have questions, concerns or feedback about my experience?

This research has been reviewed and approved by an IRB within the Human Research Protections Program (HRPP). To share feedback privately with the HRPP about your research experience, call the Research Participants' Advocate Line at <u>612-625-1650</u> (Toll Free: 1-888-224-8636) or go to <u>z.umn.edu/participants</u>. You are encouraged to contact the HRPP if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

### Will I have a chance to provide feedback after the study is over?

The HRPP may ask you to complete a survey that asks about your experience as a research participant. You do not have to complete the survey if you do not want to. If you do choose to complete the survey, your responses will be anonymous.

If you are not asked to complete a survey, but you would like to share feedback, please contact the study team or the HRPP. See the "Investigator Contact Information" of this form for study team contact information and "Whom do I contact if I have questions, concerns or feedback about my experience?" of this form for HRPP contact information.

#### Will I be compensated for my participation?

If you agree to take part in this research study, we will pay you \$100 for your time and effort after you complete the follow-up interview. You can choose if you would like to have the payment mailed to you or if you would prefer to pick up the payment at the clinic.

Payment will be made using a pre-paid debit card called Greenphire ClinCard. It works like a bank debit card.


TEMPLATE LAST REVISED: 11/1/2021
Version Date: 7 January 2025

You may use this card at any store that accepts MasterCard or you can use a bank machine to remove cash. However, there may be fees drawn against the balance of the card for cash withdrawals (ATM use) and inactivity (no use for 6 months). We will give you the ClinCard Frequently Asked Questions information sheet that answers common questions about the debit card. You will also receive a cardholder agreement. Be sure to read all of this information for details about fees.

The debit card system is administered by an outside company. The company, Greenphire, and MasterCard, will be given your name, date of birth, and address. They will use this information as part of the payment process. Greenphire will only need your social security number if the payment exceeds \$599. Greenphire and MasterCard will not receive any information about your health status or the study in which you are participating.

Payment you receive as compensation for participation in research is considered taxable income. If payment to an individual equals or exceeds \$600 in any one calendar year, the University of Minnesota is required to report this information to the Internal Revenue Service (IRS). Research payments to study participants that equal or exceed \$600 during any calendar year will result in a FORM 1099 (Miscellaneous Income) being issued to you and a copy sent to the IRS.

| <b>Signatures:</b> Your signature documents your permission to take part in this research. You will be provided a copy o this signed document. | |
|---|---|
| Signature of Participant | <br>Date |
| Printed Name of Participant | |
| Signature of Person Obtaining Consent | <br>Date |
| Printed Name of Person Obtaining Consent | |

## Signature Block for Witness (if applicable):

| <b>Witness Statement:</b> The participant was unable to read or sign this consent form because of the following reason: | |
|---|---|
| $\square$ The participant is unable to read the information | |
| ☐ The participant is visually impaired | |
| $\Box$ The participant is physically unable to sign the consent form. Please describe: | |
| □ Other (please specify): | |
| Signature of Witness | Date |
| Printed Name of Witness | |